CLINICAL TRIAL: NCT05171257
Title: Quantifying Gram-negative Resistance to Empiric Therapy in the Intensive Care Unit - Repeat ExpoSure to AntimicRobial Therapy (RESTART)
Brief Title: Quantifying Gram-negative Resistance to Empiric Therapy in the Intensive Care Unit
Acronym: RESTART
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 038.PHA.2021.D
Record Dates: First submitted 2021-12-09; First posted 2021-12-28 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Gram-Negative Bacterial Infections
MeSH Terms: conditions — Gram-Negative Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- repeat group: patients receiving empiric therapy with the same IV antibiotics from prior
  Interventions: Drug: IV antibiotic treatment from prior
- change group: patients receiving differing IV antibiotics from prior
  Interventions: Drug: differing IV antibiotic treatment

INTERVENTIONS:
Drug: IV antibiotic treatment from prior — patients receiving same IV antibiotic treatment from prior
  Groups: repeat group
Drug: differing IV antibiotic treatment — patients receiving differing IV antibiotics from prior
  Groups: change group

SUMMARY:
Antimicrobial resistance is a global health emergency estimated to be responsible for 700,000 deaths per year worldwide, and it is well known that previous antibiotic exposure is the single most contributing factor. For example, the use of non-antipseudomonal agents can increase risk for any P. aeruginosa strain; however, the use of an agent with antipseudomonal activity would select for resistance to that particular antimicrobial agent or class. Demonstrated that each additional day of exposure to any antipseudomonal beta-lactam is associated with an increased risk of new resistance development.

The study seeks to determine whether the choice of empiric therapy (i.e., the same agent versus a different agent from prior antibiotic exposure) has any effect on the likelihood of in vitro activity against GN pathogens (GNPs) in a subsequent infection.

DETAILED DESCRIPTION:
Antimicrobials are the most commonly prescribed drugs in medicine, resulting in inappropriate use in approximately 50% of cases Misuse can have devastating effects through resistance development which further complicates selection of appropriate empiric antibiotics. In cases of severe illness, it is easy for clinicians to rely on broad spectrum antibiotics to cover the majority of likely pathogens when dealing with a presumed bacterial infection. However, this practice perpetuates the cycle of resistance. Inappropriate empiric therapy is associated with worse outcomes in resistant Gram-negative (GN) bacteremia and pneumonia, so clinicians should strive for targeted coverage that is specific to the pathogen of interest when possible. Johnson et al. showed that patients with recent antibiotic exposure had greater inappropriate initial antimicrobial therapy (45.4% vs. 21.2%; p < 0.001) and higher in-hospital mortality (51.3% vs. 34.0%; p < 0.001) compared with patients without recent antibiotic exposure.

The 2020 Infectious Diseases Society of America (IDSA) Guidance on the Treatment of Antimicrobial Resistant Gram-Negative Infections reports an increased risk of resistance with antibiotic exposure in the past 30 days. Additionally, expert opinion prompts consideration of empiric coverage with a GN agent from a different class that offers comparable spectrum of activity from previous exposure. The 2019 Community-acquired Pneumonia (CAP) Guidelines from the American Thoracic Society and IDSA lists prior antibiotic use in the last 90 days as a risk factor for P. aeruginosa.The 2016 Hospital-acquired and Ventilator-associated Pneumonia (HAP, VAP) Guidelines from IDSA, list antibiotic use in the past 90 days as a risk factor for P. aeruginosa and other GN organisms in HAP. Additionally, antibiotic use in the past 90 days is listed as having an association with increased risk of multi-drug resistant VAP. The CAP, HAP, and VAP Guidelines do not mention using the same versus different agent as empiric choice if previous antibiotic exposure is to an anti-pseudomonal agent.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* GNP pneumonia or bacteremia during hospital admission
* Previous IV antibiotics for at least 48 hours in the past 90 days
* Culture MIC data available

Exclusion Criteria:

* Patients with a history of isolate resistance in the previous six months to antibiotics being studied
* Patients that received antibiotics within five days prior to study inclusion
* Patients on more than one anti-pseudomonal beta-lactam antibiotics (excluding emergency department doses) during previous exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: sample size of 242 (121 patients in each group)
Sampling Method: Probability Sample
Enrollment: 304 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Rates of resistance | charts from 4/1/2017 to 3/31/2021
  Rates of resistance in patients receiving empiric therapy with the same IV antibiotics from prior (repeat group) compared to rates of resistance in patients receiving differing IV antibiotics from prior (change group)

SECONDARY OUTCOMES:
Intensive Care Unite LOS(ICU LOS) | charts from 4/1/2017 to 3/31/2021
  Intensive Care Unite LOS(ICU LOS)

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Crotty, MD, Principal Investigator — Methodist
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No